CLINICAL TRIAL: NCT06080529
Title: Metabolic Cost of Sandbag Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Dimitrios Draganidis, Assistant Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: MET-SANDBAG-UTH
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Exercise Energy Expenditure
Keywords: Anaerobic energy expenditure; Functional training; Sandbag training; Excess post-exercise oxygen consumption; Aerobic energy expenditure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30-SEC (Experimental): Participants will execute each exercise for 30 seconds
  Interventions: Other: Sandbag exercise
- 45-SEC (Experimental): Participants will execute each exercise for 45 seconds
  Interventions: Other: Sandbag exercise

INTERVENTIONS:
Other: Sandbag exercise — Both arms include an exercise intervention consisted of 8 different exercises with sandbag: (1) lateral bag drag, (2) dead bag, (3) shoulder to shoulder thruster, (4) sumo DL with pull, (5) front lunge, (6) single leg RDL, (7) reverse lunge with rotation and (8) clean

SUMMARY:
This study aims at investigating the metabolic cost of several fundamental exercises with sandbag. Sandbag training has become a popular training modality that is efficiently used to improve cardiovascular status and physical performance. Despite its widespread use and popularity the metabolic cost of exercises using sandbag remains to be elucidated. Therefore, the metabolic cost of various fundamental exercise with sandbag will be determined to aid the planning of exercise training programs.

DETAILED DESCRIPTION:
Ten healthy young adults will be assigned to this study. Participants will initially undergo a baseline assessment of their anthropometrics, body composition (by DXA), resting metabolic rate (RMR), cardiorespiratory fitness (VO2max), muscular strength [maximal strength (1RM) and muscular endurance] and functional capacity. After baseline screening, participants will execute in different days (one exercise per day) one set of each of the following 8 exercise: (1) lateral bag drag, (2) dead bag, (3) shoulder to shoulder thruster, (4) sumo DL with pull, (5) front lunge, (6) single leg RDL, (7) reverse lunge with rotation and (8) clean, in two different conditions: (i) 30 sec and (ii) 45 sec exercise duration, in a random order. Prior to each exercise resting heart rate, blood lactate concentration, oxygen consumption and rate of perceived exertion will be recorded. Heart rate and oxygen consumption (through portable gas analyzer) will be continuously monitored during the exercise and after the end of it, until the oxygen consumption reach the pre-exercise values (excess post-exercise oxygen consumption). Blood lactate and rate of perceived exertion will be reassessed post-exercise.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 35 years
* Physically active individuals
* Free of chronic diseases
* Free of musculoskeletal injuries
* Nonsmokers

Exclusion Criteria:

* Chronic disease
* Musculoskeletal injury
* Consumption of alcohol, caffeine and any type of ergogenic supplement during the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in exercise energy expenditure | At pre-exercise, during and up to 15 minutes after the exercise (a single set lasting 30 or 45 seconds)
  Total energy expenditure (kcals) during the exercise will be assessed by summing the kcals of the oxidative system, the glycolytic system and the excess post-exercise oxygen consumption.
Change in aerobic energy expenditure | At pre-exercise and during the exercise (a single set lasting 30 or 45 seconds)
  The contribution of oxidative system in exercise energy expenditure will be assessed by the change in oxygen consumption during the exercise using a portable gas analyzer
Change in anaerobic energy expenditure | At pre-exercise and post-exercise (a single set lasting 30 or 45 seconds)
  The glycolytic contribution to exercise energy expenditure will be assessed by the change in blood lactate concentration after the exercise
Change in recovery energy expenditure | At pre-exercise and up to 15 minutes after the exercise (a single set lasting 30 or 45 seconds)
  The contribution of excess post-exercise oxygen consumption in exercise energy expenditure will be assessed by the change in oxygen consumption after the exercise using a portable gas analyzer

SECONDARY OUTCOMES:
Change in blood lactate concentration | At pre-exercise and 4 minutes after the exercise session
  Blood lactate concentration will be assessed using a portable automatic analyzer
Change in heart rate | At pre-exercise, during and up to 15 minutes after the exercise session.
  Heart rate will be assessed using a wearable heart rate monitor
Change in rate of perceived exertion | At pre-exercise and post-exercise session.
  Perceived exertion will be assessed using the Borg Rating of Perceived Exertion Scale (0-10), with ''0'' indicating ''No Exertion'' and ''10'' indicating ''Maximal Exertion''.
Change in respiratory exchange ratio | At pre-exercise, during and up to 15 minutes after the exercise session.
  Respiratory exchange ratio will be assessed using a portable gas analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Draganidis, PhD, Study Director — University of Thessaly
Locations (1):
- Laboratory of Exercise Physiology, Exercise Biochemistry and Sports Nutrition, Department of Physical Education and Sport Science, University of Thessaly, Trikala, Karyes, Greece